CLINICAL TRIAL: NCT02504502
Title: Enhancing Genomic Laboratory Reports to Enhance Communication and Empower Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Marc S. Williams, Director, Genomic Medicine Institute, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2013-0594
Record Dates: First submitted 2015-07-07; First posted 2015-07-22 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2017-08

CONDITIONS: Intellectual Disability; Autism; Multiple Congenital Anomalies
Keywords: Whole Genome Sequencing; Laboratory Report; Patient Centered; Communication of Results; Patient Provider Communication
MeSH Terms: conditions — Intellectual Disability; Autistic Disorder; Abnormalities, Multiple

STUDY DESIGN:
Intervention Model Description: intervention = routine clinical care for return of results per whole genome sequencing study with enhanced genetic test results report developed through phase 1 and 2 of this study.
  Control with delayed intervention = routine clinical care for return of results per whole genome sequencing study with crossover to receipt of enhanced report upon completion of baseline and 3 month post-baseline followup surveys. Participants in this arm will complete a third survey at 3 months post receipt of enhanced report
Who Masked: Participant
Masking Description: participants do not know whether they are in the intervention (enhanced report) or control (routine clinical care with delayed access to the enhanced report) arm
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced genomic report (Experimental): routine clinical care for return of results per whole genome sequencing study with enhanced genetic test results report developed through phase 1 and 2 of this study
  Interventions: Other: enhanced genomic report
- Control with delayed access (Other): routine clinical care for return of results per whole genome sequencing study and no intervention through three months. This arm will crossover to receipt of enhanced report upon completion of baseline and 3 month post-baseline followup surveys. Participants in this arm will complete a third survey at 3 months post receipt of enhanced report
  Interventions: Other: enhanced genomic report

INTERVENTIONS:
Other: enhanced genomic report — a patient-centered version of a genomic results report delivered to patient through the electronic record portal

SUMMARY:
Current lab reports are designed to communicate results from the laboratory to the provider; they are not designed to be accessible to patients. The investigators believe that a new type of genomic test report, tailored for patient- as well as provider-use, will enable patients to have access to information they can understand allowing them to be more involved in the management of their disorders, better navigate the health care system, and make more informed decisions about their health and health care in conjunction with their providers. This approach has the potential to improve outcomes from both the patient and provider perspectives.

The investigators propose to study the research question, "Can a genomic laboratory report tailored for both providers and families of patients improve interpretation of complex results and facilitate recommended care by enhancing communication and shared decision making?"

DETAILED DESCRIPTION:
This is a mixed-methods will be conducted in multiple phases:

Phase 1: development of an enhanced genomic test result report through in-depth interviews with parents and providers

Phase 2: refine the report through parental focus groups and provider interviews and create the final report and delivery method.

Phase 3: implement the enhanced test report and evaluate the impact on patient and providers

Subjects for the study are parents of affected children enrolled in the Whole Genome Sequencing (WGS) Clinical Research Pilot Study (study within a study). All parents receive routine clinical care for WGS and clinical return of results per protocol of the WGS study.

Parents from the WGS study were invited to participate in phases 1 and 2 of this study to help design and test an enhanced genomic test report that would meet their needs for information about their child's condition and communication with providers, caregivers, teachers, and family.

This report in clinicaltrials.gov reports on phase 3 data only. The experimental design to be used for phase 3 of the project is a randomized, single-blinded pre- post-intervention trial with crossover.

According to the WGS study protocol all results of the WGS testing will be provided by a geneticist and genetic counselor at an informing session. At this session, results will be returned and explained, recommendations provided and questions answered (routine clinical care). Following this session, parents will be randomized as couples based on whether their child received a result of a causal variant or non-causal variant to receive either routine clinical care with an enhanced report (intervention arm) or routine clinical care first followed by enhanced report (control with crossover). Randomizing parents as couples is necessary as randomization at the individual level would lead to contamination and spillover if one member of the couple were in the usual care arm and the other in the intervention arm.

After routine clinical care to deliver the WGS test results and randomization, parents will be invited to participate in phase 3 to test the impact of the enhanced report on parental and provider satisfaction, communication, and knowledge. Parents will enter into phase 3 of the study (experimental design) by completing baseline surveys. Upon completion of baseline surveys, parents will be provided the enhanced report (intervention) or another copy of their standard lab report (control with crossover).

All parents will be surveyed at 3 months. Parents in the control with crossover arm will be provided the enhanced report at this time and sent another survey 3 month post enhanced report (6 month post baseline). Standard, validated, survey instruments will be utilized for the baseline and follow-up surveys; therefore, it is possible that important differences between the routine clinical care with crossover and intervention arms could be missed. To insure capture of all important differences and all impact of the enhanced genomic test result report, additional in-depth qualitative interviews will take place after the final survey post enhanced report is administered.

ELIGIBILITY:
Inclusion Criteria:

* Research participants who are consented to participate in the WGS Study (#2012-0187).
* Providers who have referred participants to the WGS Study (#2012-0187) and who have participated in the WGS genomic medicine workgroup or who have participated in the WGS Program Oversight Committee.

Exclusion Criteria:

* Participants who are not consented to participate in the WGS Study (#2012-0187)
* Providers who have not referred patients to the WGS Study (#2012-0187).
* Providers who have not had a relationship with the oversight of the WGS study (#2012- 0187).

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc S Williams, MD, Principal Investigator — Geisinger Genomic Medicine Institute

REFERENCES:
- [Background] Scriver CR, Neal JL, Saginur R, Clow A. The frequency of genetic disease and congenital malformation among patients in a pediatric hospital. Can Med Assoc J. 1973 May 5;108(9):1111-5. PMID 4704890
- [Background] Wilson J. Acknowledging the expertise of patients and their organisations. BMJ. 1999 Sep 18;319(7212):771-4. doi: 10.1136/bmj.319.7212.771. No abstract available. PMID 10488011
- [Background] Levy HP, LoPresti L, Seibert DC. Twenty questions in genetic medicine--an assessment of World Wide Web databases for genetics information at the point of care. Genet Med. 2008 Sep;10(9):659-67. doi: 10.1097/gim.0b013e318180639d. PMID 18978677
- [Background] Morgan MA, Driscoll DA, Zinberg S, Schulkin J, Mennuti MT. Impact of self-reported familiarity with guidelines for cystic fibrosis carrier screening. Obstet Gynecol. 2005 Jun;105(6):1355-61. doi: 10.1097/01.AOG.0000163251.54416.a6. PMID 15932829
- [Background] Giardiello FM, Brensinger JD, Petersen GM, Luce MC, Hylind LM, Bacon JA, Booker SV, Parker RD, Hamilton SR. The use and interpretation of commercial APC gene testing for familial adenomatous polyposis. N Engl J Med. 1997 Mar 20;336(12):823-7. doi: 10.1056/NEJM199703203361202. PMID 9062090
- [Background] Sandhaus LM, Singer ME, Dawson NV, Wiesner GL. Reporting BRCA test results to primary care physicians. Genet Med. 2001 Sep-Oct;3(5):327-34. doi: 10.1097/00125817-200109000-00001. PMID 11545685
- [Background] Bloom BS. Effects of continuing medical education on improving physician clinical care and patient health: a review of systematic reviews. Int J Technol Assess Health Care. 2005 Summer;21(3):380-5. doi: 10.1017/s026646230505049x. PMID 16110718
- [Background] Hammond EH, Flinner RL. Clinically relevant breast cancer reporting: using process measures to improve anatomic pathology reporting. Arch Pathol Lab Med. 1997 Nov;121(11):1171-5. PMID 9372744
- [Background] Laposata ME, Laposata M, Van Cott EM, Buchner DS, Kashalo MS, Dighe AS. Physician survey of a laboratory medicine interpretive service and evaluation of the influence of interpretations on laboratory test ordering. Arch Pathol Lab Med. 2004 Dec;128(12):1424-7. doi: 10.5858/2004-128-1424-PSOALM. PMID 15578888
- [Background] Lubin IM, McGovern MM, Gibson Z, Gross SJ, Lyon E, Pagon RA, Pratt VM, Rashid J, Shaw C, Stoddard L, Trotter TL, Williams MS, Amos Wilson J, Pass K. Clinician perspectives about molecular genetic testing for heritable conditions and development of a clinician-friendly laboratory report. J Mol Diagn. 2009 Mar;11(2):162-71. doi: 10.2353/jmoldx.2009.080130. Epub 2009 Feb 5. PMID 19197001
- [Background] Scheuner MT, Hilborne L, Brown J, Lubin IM; members of the RAND Molecular Genetic Test Report Advisory Board. A report template for molecular genetic tests designed to improve communication between the clinician and laboratory. Genet Test Mol Biomarkers. 2012 Jul;16(7):761-9. doi: 10.1089/gtmb.2011.0328. Epub 2012 Jun 25. PMID 22731646
- [Background] Scheuner MT, Edelen MO, Hilborne LH, Lubin IM; RAND Molecular Genetic Test Report Advisory Board. Effective communication of molecular genetic test results to primary care providers. Genet Med. 2013 Jun;15(6):444-9. doi: 10.1038/gim.2012.151. Epub 2012 Dec 6. PMID 23222660
- [Background] Lerman CE, Brody DS, Caputo GC, Smith DG, Lazaro CG, Wolfson HG. Patients' Perceived Involvement in Care Scale: relationship to attitudes about illness and medical care. J Gen Intern Med. 1990 Jan-Feb;5(1):29-33. doi: 10.1007/BF02602306. PMID 2299426
- [Background] Cella D, Hughes C, Peterman A, Chang CH, Peshkin BN, Schwartz MD, Wenzel L, Lemke A, Marcus AC, Lerman C. A brief assessment of concerns associated with genetic testing for cancer: the Multidimensional Impact of Cancer Risk Assessment (MICRA) questionnaire. Health Psychol. 2002 Nov;21(6):564-72. PMID 12433008
- [Background] Chung WW, Chen CA, Cupples LA, Roberts JS, Hiraki SC, Nair AK, Green RC, Stern RA. A new scale measuring psychologic impact of genetic susceptibility testing for Alzheimer disease. Alzheimer Dis Assoc Disord. 2009 Jan-Mar;23(1):50-6. doi: 10.1097/wad.0b013e318188429e. PMID 19266699
- [Background] Mishel MH. Parents' perception of uncertainty concerning their hospitalized child. Nurs Res. 1983 Nov-Dec;32(6):324-30. PMID 6567851
- [Background] DuBenske LL, Burke Beckjord E, Hawkins RP, Gustafson DH. Psychometric evaluation of the Health Information Orientation Scale: a brief measure for assessing health information engagement and apprehension. J Health Psychol. 2009 Sep;14(6):721-30. doi: 10.1177/1359105309338892. PMID 19687109
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Emery AEH, Rimoin DL. 1990. Principles and Practice of Medical Genetics, Second Edition. New York, Churchill Livingstone

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects participating in the whole genome sequencing study for undiagnosed developmental delay at Geisinger Health System were invited to participate.
Pre-assignment Details: parents were randomized together (e.g. parents were both randomized to the same arm).
  parents were grouped by genomic sequencing finding (causal variant found vs. non-causal variant found) prior to randomization to ensure equal number of causal variants and non-causal variants in each arm.
Groups:
- Routine Care With Delayed Access to Report: Participants will receive routine clinical care with a copy of their standard laboratory report. After completion of the 3 month survey, participants will receive the enhanced report, followed by another survey 3 months after receiving the enhanced report.
- Routine Clinical Care Plus Enhanced Genomic Report: Routine clinical care and access to the enhanced genomic lab report upon completion of the baseline survey. Participants in this arm will receive only one survey at 3 months post enhanced report.
Period: Routine Care vs. Enhanced Report
Arm/Group | Routine Care With Delayed Access to Report | Routine Clinical Care Plus Enhanced Genomic Report
Started | 24 | 28
Completed | 20 | 21
Not Completed | 4 | 7
Not completed — Lost to Follow-up | 4 | 7
Period: Crossover to Enhanced Report
Arm/Group | Routine Care With Delayed Access to Report | Routine Clinical Care Plus Enhanced Genomic Report
Started | 20 | 0 (The enhanced report arm was completed in first period and does not carry forward to period 2.)
Completed | 15 | 0 (the enhanced report arm was completed in first period and does not carry forward to period 2)
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control With Delayed Access: Those resulting in variants of significance will receive routine clinical care and receive the enhanced genomic report after returning 3 month survey.
  Routine Clinical Care: Participants will receive routine clinical care. After returning the 3 month survey the participants will also receive the enhanced genomic report.
- Enhanced Genomic Report: Those resulting in variants of significance will received routine clinical care and access to the enhanced genomic lab report.
  Enhanced Genomic Report: Routine clinical care vs. enhanced genomic report
- Total: Total of all reporting groups
Arm/Group | Control With Delayed Access | Enhanced Genomic Report | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 28 | 52
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 23 | 26 | 49
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 23 | 26 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 28 | 52
Child's WGS Result [Count of Participants; unit: Participants] — Child's result after Whole Genome Sequencing (WGS). Results are either Causal Variant (CV) found or non-Causal Variant (NCV) found. CV indicates a positive result for the child (a genetic cause for the developmental delay). NCV indicates results were negative (no genetic cause or diagnosis for the child after sequencing).
  Participants
    Causal Variant Result | 4 | 3 | 7
    Non-Causal Variant Result | 20 | 25 | 45
Education [Count of Participants; unit: Participants] — Highest level of education completed by participant
  Participants
    Some high school (9-12) | 4 | 0 | 4
    High school graduate or GED | 3 | 7 | 10
    Post high school training other than college | 2 | 5 | 7
    Some college | 7 | 6 | 13
    Bachelor's degree or equivalent | 3 | 6 | 9
    Master's degree | 4 | 4 | 8
    Doctor or other professional degree | 1 | 0 | 1
Income [Count of Participants; unit: Participants] — Total household income
  Participants
    Less than $15,000 | 0 | 1 | 1
    $15,000 to $29,999 | 3 | 1 | 4
    $30,000 to $44,999 | 2 | 4 | 6
    $45,000 to $59,999 | 6 | 2 | 8
    $60,000 to $89,999 | 4 | 14 | 18
    $90,000 to $149,999 | 3 | 2 | 5
    $150,000 to $199,999 | 3 | 2 | 5
    $200,000 or above | 3 | 0 | 3
    Missing | 0 | 2 | 2
Health Literacy [Count of Participants; unit: Participants] — How confident are you filling out forms by yourself?
  Participants
    Never | 1 | 0 | 1
    Occasionally | 2 | 4 | 6
    Sometimes | 5 | 4 | 9
    Often | 2 | 4 | 6
    Always | 14 | 15 | 29
    Missing | 0 | 1 | 1
Numeracy [Count of Participants; unit: Participants] — In general, how easy or hard do you find it to understand medical statistics
  Participants
    Very Easy | 5 | 6 | 11
    Easy | 13 | 12 | 25
    Hard | 6 | 9 | 15
    Very Hard | 0 | 0 | 0
    Missing | 0 | 1 | 1
Access to Child's Record [Count of Participants; unit: Participants] — How many times did you access your child's health information online through the MyGeisinger website or app in the last 12 months?
  Participants
    None | 12 | 17 | 29
    1-2 times | 2 | 2 | 4
    3-5 times | 5 | 3 | 8
    6-9 times | 0 | 2 | 2
    10 or more times | 4 | 3 | 7
    Missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With Genomic Test Report
Description: 3 questions on how helpful various parts of the test report were for parents who opened the enhanced report.
Time Frame: 3 months after receipt of enhanced report
Population: parents who opened the enhanced report per electronic confirmation. For Clinical care then enhanced report N=4 CV; 2NCV - these 2 NCV parents did not answer the survey questions about the report ("missing"). For routine care with enhanced report first N=9 NCV.
Measure: Count of Participants; unit: Participants
Groups:
- Routine Clinical Care First, Then Enhanced Report: Participants will receive routine clinical care with a copy of their standard laboratory report. After completion of the 3 month survey, participants will receive the enhanced report, followed by another survey 3 months after receiving the enhanced report.
Arm/Group | Routine Clinical Care First, Then Enhanced Report | Routine Clinical Care Plus Enhanced Genomic Report
Number analyzed (Participants) | 6 | 9
Participants
  Summary: Not Helpful | 0 | 2
  Summary: A little bit helpfu | 1 | 1
  Summary: Somewhat helpful | 1 | 1
  Summary: Quite a bit helpful | 2 | 3
  Summary: Very helpful | 0 | 1
  Summary: Missing | 2 | 1
  Detailed Explanation: Not Helpful | 0 | 2
  Detailed Explanation: A little bit helpfu | 1 | 1
  Detailed Explanation: Somewhat helpful | 1 | 1
  Detailed Explanation: Quite a bit helpful | 2 | 1
  Detailed Explanation: Very helpful | 0 | 3
  Detailed Explanation: Missing | 2 | 1
  Care Instructions: Not Helpful | 0 | 4
  Care Instructions: A little bit helpfu | 2 | 1
  Care Instructions: Somewhat helpful | 1 | 2
  Care Instructions: Quite a bit helpful | 1 | 0
  Care Instructions: Very helpful | 0 | 1
  Care Instructions: Missing | 2 | 1

ADVERSE EVENTS:
Time Frame: study duration, up to 6 months post receipt of enhanced genomic results report
Arm/Group | Routine Clinical Care First, Then Enhanced Report | Routine Clinical Care Plus Enhanced Genomic Report
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/28
Other Adverse Events (participants affected / at risk) | 0/24 | 0/28

LIMITATIONS AND CAVEATS:
Fewer parents than expected received a causal variant result for their child's condition. Qualitative data indicate that parents without a causal variant did not feel need to open the enhanced report and did not find additional information helpful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes